CLINICAL TRIAL: NCT03986814
Title: Exposure to Air Pollutants and Green Space: Implications for the Gut Microbiome and Metabolome in Young Adults Living in Denver, Colorado
Brief Title: Environmental Health Effects on Your Physiology
Acronym: HYPHY
Status: Completed | Type: Observational
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Tanya Alderete, Assistant Professor, University of Colorado, Boulder
Other Study IDs: 19-0201
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and fecal samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the associations between exposure to air pollutants, green space, and the gut microbiome and metabolome.

DETAILED DESCRIPTION:
A rapidly evolving field of study suggests a link between the gut microbiome and fecal metabolome with obesity. Recent studies show that environmental exposures, such as ambient air pollution (AAP) exposure can affect gut bacteria and modify risk for obesity. Additionally, proximity to green space has been shown to reduce exposure to air pollutants and increase gut microbial diversity. The investigator's preliminary work has shown that near-roadway air pollution exposure was positively correlated with gut microbial taxa that have been linked with obesity. These findings suggest that air pollution exposure may increase susceptibility to obesity through alterations in the composition and function of the gut microbiome. Despite this, no studies have systematically examined the impact of air pollutants and green space on the gut microbiome and metabolome among adolescents. The overall goal of this research is to determine whether exposure to air pollutants and/or green space affect the gut microbiome and metabolome in young adults residing in Denver, Colorado. This study will examine residential-based estimates of air pollution exposure and green space and also perform detailed gut microbial and metabolite profiling in 100 adolescent and young adults.

ELIGIBILITY:
Inclusion Criteria:

* The participant population includes young adults (18-25 years of age) who live in Denver, Colorado.

Exclusion Criteria:

* Exclusion criteria include physical, mental, or cognitive disability that prevents participation
* Current incarceration
* Antibiotic usage in the previous month
* Pregnant or nursing
* Non-English speaking
* Any medical conditions known to affect body composition, insulin secretion, or the gut microbiota (i.e., type 1 or 2 diabetes, intestinal bowel disease, Crohn's Disease, kidney disease, heart disease, autoimmune disease).

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Young adults from Denver, Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-02-13 (Actual)

PRIMARY OUTCOMES:
Gut Microbiome | Measured once at baseline visit date
  16S rRNA and Shotgun Sequencing
Fecal Metabolome | Measured once at baseline visit date
  Targeted and/or Un-targeted Metabolomics
Body mass index (BMI) | Measured once at baseline visit date
  Weight and height will be combined to report BMI in kg/m^2
Body Composition | Measured once at baseline visit date
  Waist and hip measurements will be taken

SECONDARY OUTCOMES:
Air Pollution | One year before baseline visit date
  Modeled residential exposure to air pollution
Green Space | One year before baseline visit date
  Modeled residential exposure to green space
Serum Metabolome | Measured once at baseline visit date
  Targeted and/or Un-targeted Metabolomics
Diet | Measured once at baseline
  Automated Self-Administered 24-Hour (ASA24)
Physical Activity | Measured once at baseline
  International Physical Activity Questionnaire
Fasting Glucose | Measured once at baseline
  Fasting Glucose (mg/dl)
Fasting Insulin | Measured once at baseline
  Fasting insulin (uU/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Research Center, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No